CLINICAL TRIAL: NCT00472784
Title: Quantitative and Qualitative Changes in Neural Efferent Receptors, Collagen and Smooth Muscle Content in the Bladder, Following Spinal Cord Injury (SCI) in Humans
Brief Title: Quantitative and Qualitative Changes in Neural Efferent Receptors
Status: Withdrawn | Type: Observational
Why Stopped: Study no longer being conducted.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Christopher Patrick Smith, Associate Professor, Baylor College of Medicine
Other Study IDs: H-6079
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Spinal Cord Injury; Bladder Dysfunction
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
OBJECTIVE: 1. To study tissues from spinal cord injured patients with noncompliant bladders as well as neurologically intact patients with normal bladder compliance, analyzing both quantitative and qualitative neural efferent receptors, collagen, and smooth muscle contents, using RT-PCR and electron microscopy. 2. To explore the possible shift in bladder neural architecture after SCI from beta to alpha-adrenergic receptors.

RESEARCH DESIGN: 25 spinal cord injury patients who underwent cystoscopic procedures will be included in this study. 25 control patients without spinal cord injury and already scheduled for urologic procedures will also be included in this study.

METHODOLOGY: Study patients will undergo flexible or rigid cystoscopy as well as selective cold cup biopsies of the posterior and lateral walls, and trigonal area of the bladder. Control patents will undergo cystoscopy and selected bladder biopsies preceding their scheduled urologic procedures. Tissue samples will be frozen for later EM and RT-PCR analysis of collagen, smooth muscle, and efferent adrenergic receptor content and subtype. Hemostasis will be achieved with a cautery electrode. Criteria of exclusion include active urinary tract infection identified by preoperative urinalysis, or the presence of suspicious lesions seen during cystoscopy. Suspicious areas will be biopsied and the patient will be excluded from the study.

Subjects will be given a preoperative dose of Rocephin 1g IM as well as a postoperative 3-day course of Cipro 500 mg BID. Control patients will be given standard perioperative prophylactic/empiric therapy as indicated for their urologic procedure. Patients will be followed in 1-2 weeks to evaluate their postoperative course.

FINDINGS: Total number of subjects enrolled: 43. 12-03: To date we have not encountered any problems with the study and health wise the subjects have done fine. No adverse events have been reported. Preliminary Results: The tissue is currently being analyzed - mRNA by microchip analysis and the data is still being worked on to look for correlations in genes up or down regulation versus the morphological EM findings previously reported.

DETAILED DESCRIPTION:
Twenty-five (25) spinal cord injury patients, as part of their annual cystoscopic screening for squamous cell carcinoma, will be included in this study. Approximately twenty-five (25) control patients without spinal cord injury and already scheduled for cystoscopic procedures (transurethral resection of the prostate TURP for benign prostatic hyperplasia BPH, transurethral resection of low-grade superficial bladder tumor TURBT, or lithotripsy of urinary stones) will be included in this study. Enrollment of additional patients is necessary to increase the statistical power to demonstrate significant difference between the study and control groups. Preliminary results revealed that electron microscopy was accurate at differentiating neurogenic detrusor muscle from normal. There was a strong trend towards increased type I/type III collagen expression in SCI patients versus normal, but recruitment of more patients is necessary to demonstrate unequivocally a statistical difference.

Patients will undergo flexible or rigid cystoscopy as well as selective cold cup biopsies of the posterior and lateral walls, and trigonal area of the bladder. Bladder mapping (diagram attached) will be performed to document specific areas biopsied. Tissue samples will be frozen for later RT-PCR analysis of collagen, smooth muscle, and efferent adrenergic receptor content and subtype. No anesthesia will be required in the SCI study patients. Control group patients will undergo anesthesia as indicated by their TURP or cystoscopic procedure.

Hemostasis will be achieved with a cautery electrode. Criteria for exclusion include active urinary tract infection identified by preoperative urinalysis. Patients with low-grade superficial bladder tumor, which has a classic cystoscopic appearance, is no longer excluded from the study since directed cold cup bladder biopsies at sites away from the visible tumor (obtained from the posterior, both lateral walls, as well as the trigone of the bladder) is now considered standard of care to rule out occult carcinoma-in-situ (CIS).

Prophylactic perioperative antibiotics will be employed. Patients will be followed in 1-2 weeks to evaluate their postoperative course.

Annual cystoscopy in spinal cord injured patients to screen for squamous cell carcinoma as well as preoperative cystoscopy in TURP, TURBT, and lithotripsy candidates is considered standard clinical care.

Selective bladder biopsies of normal appearing bladder mucosa and muscle are included as part of this study protocol.

Study patients will be given a preoperative dose of Rocephin 1 gm IM as well as a postoperative 3-day course of Cipro 500mg BD. Control patients will be given standard perioperative prophylactic/empiric therapy as indicated for their scheduled cystoscopic procedures.

Study patients will be scheduled for two visits. The first visit as part of their annual exam, to include cystoscopy, and bladder biopsies, will last approximately one hour. The second visit, two weeks later, will examine the patient's postoperative course. This visit will last approximately 15 minutes. Control patients will undergo cystoscopy and selected bladder biopsies preceding their already scheduled cystoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Informed and consenting adult VA patients with either:

  1. spinal cord injury and documented noncompliant bladders by urodynamics (n=20,
  2. men with normal bladder compliance (n=5, >20cc/cm H20) scheduled for TURP or TURBT or lithotripsy

Exclusion Criteria:

* Patients with active urinary infections

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Spinal cord injury Bladder dysfunction
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 1998-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The tissue is currently being analyzed - mRNA by microchip analysis and the data is still being worked on to look for correlations in genes up or down regulation versus the morphological EM findings previously reported. | 9 years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P. Smith, M.D., Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor College of Medicine - Scott Department of Urology, Houston, Texas
  - Michael E. DeBakey Veteran's Affairs Medcial Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No